CLINICAL TRIAL: NCT07349199
Title: Adherence to Clinical Guidelines on Perioperative Diabetes Care in Hospitalised Patients. A Retrospective Cohort Study.
Brief Title: Adherence to Clinical Guidelines on Perioperative Diabetes Care
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Steno Diabetes Center Copenhagen (Other); Steno Diabetes Center Sjaelland (Other Government); Rigshospitalet, Denmark (Other); Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Casper Pedersen, MD, PhD student, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: R-25014694
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Perioperative Medicine; Diabetes (DM); Diabetes Mellitus
Keywords: Diabetic care; Perioperative medicine; Guidelines adherence; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with type 1 or type 2 diabetes mellitus undergoing non-cardiac surgery >1 hour duration

SUMMARY:
Patients who undergo major surgery face a 15-30% risk of serious adverse events, including a 1-5% mortality risk in the first month after surgery. For patients with diabetes, the risk is even greater, and it is often aggravated by complications associated with hyper- and hypoglycaemia. Complications, such as wound infections, cardiovascular, and neurological events, not only affect patients negatively, but it challenges health care systems due to prolonged length of stays and increased need of care post-discharge.

Several factors make it particularly difficult to establish glycaemic control and stable blood sugar in patients with diabetes. Patients' usual glucose-lowering medications are often paused, and fasting is required at least six hours prior to the operation. Surgery induces a post-surgical stress response that may include both stress-hyperglycaemia and reduced gastrointestinal function. Furthermore, a patient's usual symptoms of hyper- and hypoglycaemia may be altered due to the anaesthetics.

The existing guidelines on perioperative diabetic care include recommendations on treatment and glucose monitoring from the preoperative fasting period to the postoperative phase where oral intake of food and drinks can be resumed. Intravenous glucose-insulin infusions are used during preoperative fasting, intraoperatively and postoperatively until patients can resume oral intake of food and drinks. After this, subcutaneous insulin administrations following the sliding scale insulin regimen are administered to the patients to treat hyperglycaemia and supplemental glucose (perorally or intravenously) in case of hypoglycaemia. The blood sugar levels are monitored via point-of-care (POC) blood glucose tests every hour during glucose-insulin infusions and four to six times daily in the postoperative period.

In spite of these guidelines, prospective studies have shown that blood glucose levels are outside the normal range in 40-60% of the time following major surgery, and usually due to hyperglycaemia.

In this registry study, we investigated how guidelines for perioperative diabetes care were implemented in Danish hospitals from 2017-2023. The primary hypothesis was that, in the 20% of cases with detected hyperglycaemia, insufficient insulin was provided thus not following exiting guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years of age or older
* Type 1 or Type 2 diabetes mellitus requiring glucose-lowering medication
* Non-cardiac surgery lasting min. 1hour

Exclusion Criteria:

* Patients using insulin pump
* Planned surgery for pancreatectomy (complete or partial)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population consists of patients living with diabetes mellitus requiring glucose-lowering medication who undergo surgery in the period from Janurary 1st, 2017 to Janurary 1st, 2023 across hospitals in two regions of Denmark - the Capital Region and the Zealand Region of Denmark .
Sampling Method: Non-Probability Sample
Enrollment: 22000 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of correct insulin dose administration for hyperglycaemia | Following surgery, from the patient arrive at the surgical ward until discharge from the surgical ward, up to 30 days postoperative
  The proportion of hyperglycaemic events in which the recommended insulin dose, according to the interregional guideline, is administered. Correct dosing is defined as administration of the guideline-recommended dose of rapid-acting insulin (international units [IU], whole numbers) from 15 min. prior to 1 hour after detection of hyperglycaemia.

SECONDARY OUTCOMES:
Frequency of missing insulin administration for hyperglycaemia | Following surgery, from the patient arrive at the surgical ward until discharge from the surgical ward, up to 30 days postoperative
  The proportion of hyperglycaemic events in which the recommended insulin dose, according to the interregional guideline, is NOT administered. Correct dosing is defined as administration of the guideline-recommended dose of rapid-acting insulin (international units [IU], whole numbers) from 15 min. prior to 1 hour after detection of hyperglycaemia.
Frequency of insufficient insulin dose administration for hyperglycaemia | Following surgery, from the patient arrive at the surgical ward until discharge from the surgical ward, up to 30 days postoperative
  The proportion of hyperglycaemic events in which a lower insulin dose than the recommended insulin dose, according to the interregional guideline, is administered. Correct dosing is defined as administration of the guideline-recommended dose of rapid-acting insulin (international units [IU], whole numbers) from 15 min. prior to 1 hour after detection of hyperglycaemia.

CONTACTS AND LOCATIONS:
Overall Officials: Christian S Meyhoff, Study Chair — Department of Anaesthesia and Intensive Care, Bispebjerg and Frederiksberg Hospital, Copenhagen, Denmark
Locations (1):
- Copenhagen University Hospital, Bispebjerg and Frederiksberg, Copenhagen, Denmark, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.